CLINICAL TRIAL: NCT06135363
Title: A Single-center, Open Label Study to Evaluate the Safety，Tolerability and Pharmacokinetics of Multiple Administration of Sufenidone (SC1011) Tablets in Healthy Adult Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetic Study of SC1011 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JYP1011M102
Record Dates: First submitted 2023-11-04; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Lung Diseases; Respiratory Tract Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple doses SC1011 300mg（A1） (Experimental): Drug: SC1011 tablet, SC1011-matching placebo tablet; Treatment: Food intake prior to dosing
  Interventions: Drug: SC1011; Drug: Placebo tablet
- Multiple doses SC1011 400mg（A2） (Experimental): Drug: SC1011 tablet; Treatment: Food intake prior to dosing
  Interventions: Drug: SC1011; Drug: Placebo tablet

INTERVENTIONS:
Drug: SC1011 — SC1011 tablet
  Other Names: experimental drug group
Drug: Placebo tablet — SC1011-matching placebo tablet
  Other Names: Control Group

SUMMARY:
The goal of this clinical trial is to learn about the safety, tolerability and pharmacokinetic profiles of SC1011 in healthy conditions. The main questions it aims to answer are: Safety and tolerability profiles in healthy subjects and pharmacokinetic profiles in healthy subjects. Participants will complete the study including screening period, dosing period, and observation period. Investigators will compare the inhibitory activity of SC1011 tablets with pirfenidone capsules against the same biomarkers(e.g. blood TNFα) to see if they are different between the two drugs.

DETAILED DESCRIPTION:
This is a single-center, open label study to evaluate the safety，tolerability and pharmacokinetics of multiple administration of Sufenidone (SC1011) tablets conducted in 2 groups.

Eight subjects were enrolled in the sulforaphane 300 mg group and each subject was administered once within half an hour after breakfast on day 1, twice daily on days 2-6 and once within half an hour after breakfast on day 7 .

Eight subjects were enrolled in the sulforaphane 400 mg group and each subject was administered for 7 consecutive days, with dosing consisting of one dose within half an hour after breakfast on day 1, twice daily on days 2-6, and once within half an hour after breakfast on day 7.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of any race, between 18 and 45 years of age, inclusive, at Screening.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at Screening.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and/or Check-in as assessed by the Investigator.
* Females will be nonpregnant and nonlactating. Females of childbearing potential and male subjects will agree to use contraception.
* Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance.
* Alcohol consumption of > 21 units per week for males and > 14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL wine), or a positive alcohol breath test at Check-in.
* Any screening laboratory or ECG results are not within the normal reference range and are considered clinically significant.
* Participants who participated in other clinical trials within 3 months prior to administration.
* Blood donation or blood loss exceeding 400 mL within 2 months prior to administration.
* Participants who smoked, drank alcohol, tea, food or drink containing xanthine or caffeine, or had strenuous exercise, or had other factors affecting drug absorption, distribution, metabolism and excretion 2 days before drug administration.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-01-14 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events related drug. | From baseline to 7 days
  Adverse events are coded according to the ICH Medical Dictionary of Regulatory Activities (MedDRA 24.0 or above). ADR: Adverse events that are "definitely related, probably related, or undetermined" in relation to the investigational drug.

SECONDARY OUTCOMES:
Geometric Mean of Maximum Observed Plasma Concentration of SC1011 | From baseline to 7 days
  Area under the plasma concentration-time curve (AUC) from time zero to infinity of SC1011

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No